CLINICAL TRIAL: NCT04041037
Title: The Management of Pilonidal Wounds With ACell MicroMatrix® and Cytal® Wound Matrix: A Case Series
Status: Terminated | Type: Observational
Why Stopped: Sponsor Decision
Sponsor: Integra LifeSciences Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: CR2018-001
Record Dates: First submitted 2019-07-30; First posted 2019-08-01 (Actual); Results first posted 2020-07-15 (Actual); Last update posted 2021-04-20 (Actual); Status verified 2021-03

CONDITIONS: Pilonidal Disease
Keywords: ACell; ACell MicroMatrix®; ACell Cytal® Wound Matrix; Urinary Bladder Matrix

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: Wound Sheet Matrix 2-Layer and Powder Urinary Bladder Matrix — Porcine-derived extracellular matrix will be used in powder and 2-Layer wound sheet form in masses up to 1000 mg. Each product is intended for a one-time use only.

SUMMARY:
A case series involving the concomitant use of MicroMatrix® and Cytal® Wound Matrix 2-Layer with standard of care negative pressure wound therapy (NPWT) during the management of pilonidal wound healing.

DETAILED DESCRIPTION:
This is a prospective case series examining the concomitant use of MicroMatrix® and Cytal® Wound Matrix 2-Layer with standard of care negative pressure wound therapy (NPWT) during the management of pilonidal wound healing. Wound healing will be evaluated at 2 weeks, 6 weeks, and 3 months. If subjects heal prior to the 3 month visit, wound healing will be documented at that visit. A maximum of ten subjects will be included in this series.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has a clinical diagnosis of pilonidal disease.
2. Subject is being scheduled for surgical excision of pilonidal disease.
3. Subject is at least 18 years of age.
4. Subject is willing and able to adhere to protocol requirements and agrees to participate in the study program and comply with the study follow-up regimen.
5. Subject is willing to provide written informed consent.

Exclusion Criteria:

1. Subject has a known allergy to porcine-based materials.
2. Subject is pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be selected from the medical offices of the Principal Investigator, Dr. Massarotti, and CO-Investigator, Dr. Chudzinski.
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2019-03-26 (Actual); Primary Completion 2019-08-30 (Actual); Study Completion 2019-11-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Haane Massarotti, MD, Principal Investigator — Florida Hospital Tampa
Locations (1):
- AdventHealth Tampa, Tampa, Florida, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- All Participants: Participants received MicroMatrix and Cytal Wound Matrix 2-layer in addition to Negative Pressure Wound Therapy on their pilonidal wounds.
Period: Overall Study
Arm/Group | All Participants
Started | 2
Completed | 2
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: The study was terminated by Sponsor; no data outcome analyses were conducted.
Groups:
- All Participants: All participants received MicroMatrix and Cytal Wound Matrix 2-layer in addition to Negative Pressure Wound Therapy on their pilonidal wounds.
Arm/Group | All Participants
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Rate of Wound Closure
Description: The study was terminated by Sponsor; no outcome measure data analyses were conducted.
Time Frame: Up to 3 month visit
Population: Data was collected from the two participants in the study however, rate of wound closure was not analyzed due to an extremely small sample size and study termination by Sponsor.
Arm/Group | All Participants
Number analyzed (Participants) | 0

2. Other Pre Specified Outcome: Visual Analogue Scale (VAS) for Pain
Description: The study was terminated by Sponsor; no outcome measure data analyses were conducted.
Time Frame: Up to 3 month visit
Population: The study was terminated by sponsor; no outcome measure data analyses were conducted. The Investigator was not able to achieve the enrollment goal to allow for data analyses.
Arm/Group | All Participants
Number analyzed (Participants) | 0

3. Other Pre Specified Outcome: Katz Index of Independence in Activities of Daily Living (KATZ ADL)
Description: The study was terminated by Sponsor; no outcome measure data analyses were conducted.
Time Frame: Up to 3 month visit
Population: as for outcome 2
Arm/Group | All Participants
Number analyzed (Participants) | 0

4. Other Pre Specified Outcome: Wound Related Adverse Events
Description: Number and type of wound related adverse events as recorded on adverse event case report forms
Time Frame: Up to 3 month visit
Population: as for outcome 2
Arm/Group | All Participants
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 5 months
Groups:
- All Participants: All participants received MicroMatrix and Cytal Wound Matrix 2-layer in addition to standard of care Negative Pressure Wound Therapy on their pilonidal wounds.
Arm/Group | All Participants
All-Cause Mortality (participants affected / at risk) | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 1/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Participants (N=2)
Bacterial Infection (Infections and infestations) | 1 (1) — The Subject presented with surgical site infection at their 6 weeks visit.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-02): https://cdn.clinicaltrials.gov/large-docs/37/NCT04041037/Prot_SAP_000.pdf